CLINICAL TRIAL: NCT06944561
Title: Improved Diagnostics for Paediatric Tuberculosis
Acronym: TiKa-PAEDTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JRES: 2020.0261
Record Dates: First submitted 2025-01-31; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis
Keywords: paediatric; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paediatric participants in the trial (Experimental): Any patient under the age of 21 years with the following diagnosis for whom informed consent could be obtained was offered to be included in the trial.
  * Latent tuberculosis
  * Culture confirmed Tuberculosis
  * Clinically suspected Tuberculosis
  Interventions: Diagnostic Test: Culture and identify Mycobacterium tuberculosis from patient faeces

INTERVENTIONS:
Diagnostic Test: Culture and identify Mycobacterium tuberculosis from patient faeces — When faecal samples have been identified only by a pseudo-anonymised label they will be transferred to the designated secure collection point (Vaccine Institute). Professor Tim Bull will then be informed of their availability and will collect and transport to the research laboratory, located in the same building, making a log of all samples received. All samples will then be processed by the research laboratory as defined in the sample processing protocol. Culture result data will be obtained and stored on a secure password protected PC Excel file for collation and archiving by the chief analyst.
  Other Names: Diagnostic; Culture

SUMMARY:
Improved diagnostics for paediatric Tuberculosis

DETAILED DESCRIPTION:
Research Question: To test the feasibility of TiKa system to reliably detect Mycobacterium tuberculosis in faeces of paediatric patients with Tuberculosis Study Design: Non-randomised diagnostic proof of concept feasibility study Study Participants: Patients with or suspected to have Tuberculosis

ELIGIBILITY:
Inclusion Criteria:

* Any patient under the age of 21 years with the following diagnosis for whom informed consent can be obtained will be offered to be included in the trial.

  * Latent tuberculosis
  * Culture confirmed Tuberculosis
  * Clinically suspected Tuberculosis

Exclusion Criteria:

* Any patient over 21
* Any child or adult/guardian unable to give informed consent
* Any persons under detention will not be included.
* Any patient who is unable to give a sample.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
To quantitate the speed of new culture method (TiKa) and compare its efficacy with conventional systems in detecting Mycobacterium tuberculosis in the faeces of paediatric patients with tuberculosis. | 2 years
  Samples will only include faeces (up to 10g) obtained once from outpatients and up to once per day for in-patients.
  Faecal samples will be collected and placed into a routine sterile stool collection kit, labelled with a unique identifier allocated from its associated CRF and safe transport arranged to deliver the specimen to the research laboratory. On arrival all samples will be logged and a record kept in a secure locked site by a member of the research team.

CONTACTS AND LOCATIONS:
Locations (1):
- CIU Office, St George's NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Analysed final data for release and publication will be retained and shared according to SGUL data management policy (http://www.sgul.ac.uk/images/about/Policies/SGUL_RDM_Policy_May_2016.pdf) within the SGUL data management repository. This data will not include personal identifiers and will pose no risk to ethical considerations.
  The scope and nature of the data for processing will include. 1. Paediatric patient clinical history including age, sex and results of any routine investigations related to obtaining a diagnosis of tuberculosis. 2. Sample description, sample positivity (isolation of Mycobacterium tuberculosis achieved), sample infectious load and time to positivity. All data will be kept for 5 years post study termination/end.